CLINICAL TRIAL: NCT03403361
Title: A Virtual Clinical Trial to Assess the Impact of Dual-Energy CT on Plan Quality, Dose-delivery Accuracy, and Simulated Outcomes of Patients Treated With Proton or Photon Therapy
Brief Title: Dual-Energy CT on Plan Quality, Dose-delivery Accuracy, and Simulated Outcomes of Patients Treated With Proton or Photon Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201711149; 1R01CA212638 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Brain Cancer; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dual-Energy CT scan (Experimental): Patients enrolling in this study will undergo additional sequential DECT scan in addition to their routine SECT or DECT scan.
  Interventions: Device: Siemens Somatom Definition Edge; Device: Philips Brilliance Big Bore CT/simulator

INTERVENTIONS:
Device: Siemens Somatom Definition Edge — In addition to acquiring medically-routine datasets, each patient subject will be scanned sequentially at two or three different beam energies (80 or 90 kVp, 100 kVp, 120 kVp, and 140 kVp) as part of this research study.
Device: Philips Brilliance Big Bore CT/simulator — In addition to acquiring medically-routine datasets, each patient subject will be scanned sequentially at two or three different beam energies (80 or 90 kVp, 100 kVp, 120 kVp, and 140 kVp) as part of this research study.

SUMMARY:
The aim of this protocol is to refine the accuracy of proton beam therapy (PT) by the use of dual energy computed tomography (DECT), in conjunction with novel iterative image reconstruction algorithms, to more precisely determine the tissue properties through which the proton beam path travels.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Diagnosis of histologically proven primary or metastatic cancer requiring thoracic radiation therapy OR radiation therapy to the head and neck or brain
* At least 18 years of age.
* Planning to undergo proton or photon beam radiation therapy as part of the clinical management of the diagnosed cancer.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Implanted metallic objects in the region to be scanned excepting dental prostheses
* IV or oral contrast medium within 24 hours prior to DECT image acqusition
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dual-Energy CT Scan
Started | 36
Completed | 20
Not Completed | 16
Not completed — Not imaged due to issues during the pandemic | 16

BASELINE CHARACTERISTICS:
Arm/Group | Dual-Energy CT Scan
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 66.5 [22 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Dose Difference in 99% Planning Target Volume (PTV) Coverage Between Single Energy CT and Dual Energy CT
Time Frame: Day 1
Population: 16 participants did not have imaging due to staffing changes and lack of communication during the pandemic.
Measure: Mean (Standard Deviation); unit: percentage relative to prescribed dose
Arm/Group | Dual-Energy CT Scan
Number analyzed (Participants) | 20
percentage relative to prescribed dose
  Head and Neck Patients: number analyzed (Participants) | 9
  Head and Neck Patients | 0.9 (1.8)
  Lung Patients: number analyzed (Participants) | 11
  Lung Patients | 1.0 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were followed for 1 day.
Arm/Group | Dual-Energy CT Scan
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03403361/Prot_SAP_000.pdf